CLINICAL TRIAL: NCT00916370
Title: SPIRIT PRIME Clinical Trial.
Acronym: SPIRIT PRIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-373
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; stents; Angioplasty; myocardial ischemia; coronary artery stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Long lesion
MeSH Terms: conditions — Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Core size registry (CSR) (Experimental): Core size indicates the range of diameters of the stents used.
  Interventions: Device: Core size Xience Prime
- Long lesion registry (LLR) (Experimental): Use of long lesion stents.
  Interventions: Device: Xience Prime Long Lesion (LL)

INTERVENTIONS:
Device: Core size Xience Prime — Core size includes a range of stent sizes.
  Arms: Core size registry (CSR)
Device: Xience Prime Long Lesion (LL) — Long lesion stent sizes include a range of sizes.
  Arms: Long lesion registry (LLR)

SUMMARY:
To evaluate the safety and effectiveness of the XIENCE PRIME and XIENCE PRIME Long Lesion (LL) Everolimus Eluting Coronary Stent System (EECSS) in improving coronary luminal diameter in subjects with symptomatic heart disease due to a maximum of two de novo native coronary artery lesions, each in a different epicardial vessel.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedure, per site requirements.
3. Subject must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia).
4. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Subject must agree to undergo all protocol-required follow-up procedures.
6. Subject must agree not to participate in any other clinical study for a period of one year following the index procedure.

Angiographic Inclusion Criteria

1. One or two de novo target lesions each in a different epicardial vessel.
2. If there are two target lesions, both lesions must satisfy the angiographic eligibility criteria for that registry.

   o Multiple focal de novo lesions in a target vessel that can be covered by a single stent are allowed.
3. The target lesion(s) must be located in a major artery or branch with a visually estimated diameter stenosis of ≥ 50% and < 100% with a TIMI flow of ≥ 1.
4. Target lesion(s) must be located in a native coronary artery with reference vessel diameter (RVD) by visual estimation of:

   * ≥ 2.25 mm and ≤ 4.25 mm for treatment by the core size XIENCE PRIME EECS
   * ≥ 2.5 mm and ≤ 4.25 mm for treatment by the XIENCE PRIME LL EECS
5. Target lesion(s) must be located in a native coronary artery with length by visual estimation of:

   * ≤ 22 mm for treatment by the core size XIENCE PRIME EECS
   * > 22 mm and ≤ 32 mm for treatment by the XIENCE PRIME LL EECS

Exclusion Criteria:

1. Subject has had a known diagnosis of acute myocardial infarction (AMI) preceding the index procedure (CK-MB ≥ 2 times upper limit of normal) and CK and CK-MB have not returned to within normal limits at the time of procedure.
2. The subject is currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain with ischemic ECG changes.
3. Subject has current unstable cardiac arrhythmias associated with hemodynamic instability.
4. Subject has a known left ventricular ejection fraction (LVEF) < 30% (LVEF may be obtained at the time of the index procedure if the value is unknown and if necessary).
5. Subject has received coronary brachytherapy in any epicardial vessel (target or non target).
6. Subject has received any organ transplant or is on a waiting list for any organ transplant.
7. Subject is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or within one year after the index procedure.
8. Subject is receiving or scheduled to receive planned radiotherapy to the chest/mediastinum.
9. Subject is receiving immunosuppressant therapy or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.).
10. Subject is receiving chronic anticoagulation therapy (e.g., heparin, coumadin).
11. Subject will require Low Molecular Weight Heparin (LMWH) post-procedure.
12. Subject has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
13. Elective surgery is planned within 12 months after the procedure that will require discontinuing either aspirin or clopidogrel.
14. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a white blood cell (WBC) of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis).
15. Subject has known renal insufficiency (examples being but not limited to estimated glomerular filtration rate (eGFR) < 60 ml/kg/m2, serum creatinine level ≥ 2.5 mg/dL, or on dialysis).
16. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
17. Subject has had a cerebrovascular accident/stroke or transient ischemic neurological attack (TIA) within the past six months.
18. Subject has had a significant gastro-intestinal or significant urinary bleed within the past six months.
19. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion.
20. Subject has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
21. Subject is currently participating in another clinical study that has not yet completed its primary endpoint.
22. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

Angiographic Exclusion Criteria All angiographic exclusion criteria are based on visual estimation.

1. Target lesion located within an arterial or saphenous vein graft or distal to a diseased (vessel irregularity per angiogram and > 20% stenosed lesion) arterial or saphenous vein graft.
2. Target lesion involving a bifurcation with a side branch ≥ 2 mm in diameter and/or ostial lesion > 40% stenosed or side branch requiring protection guide wire, or side branch requiring dilatation.
3. Target lesion with total occlusion (TIMI flow 0), prior to crossing with the wire.
4. Another lesion requiring revascularization is located in the same epicardial vessel of the target lesion.
5. Restenotic target lesion.
6. Aorto-ostial target lesion (within 3 mm of the aorta junction).
7. Target lesion is in a left main location.
8. Target lesion located within 2 mm of the origin of the LAD or LCX.
9. Extreme angulation (≥ 90 °) or excessive tortuosity (≥ two 45° angles) proximal to or within the lesion.
10. Heavy calcification proximal to or within the target lesion.
11. Target vessel contains thrombus as indicated in the angiographic images.
12. Target lesion has a high probability that a procedure other than pre-dilatation and stenting will be required at the time of index procedure for treatment of the target vessel (e.g. atherectomy, cutting balloon).
13. Target vessel is previously treated with any type of PCI (e.g. balloon angioplasty, stent, cutting balloon, atherectomy) < 9 months prior to index procedure.
14. Non-target vessel is previously treated with any type of PCI < 90 days prior to the index procedure.
15. Additional clinically significant lesion(s) (e.g. %DS ≥ 50%) in a target vessel or side branch for which PCI may be required < 90 days after the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Costa, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (62):
- United States (56):
  - Thomas Hospital, Fairhope, Alabama
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Mercy General Hospital, Sacramento, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - St. Vincents Medical Center, Jacksonville, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Sacred Heart Hospital of Pensicola, Pensacola, Florida
  - St. John's Hospital, Springfield, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center P.C., West Des Moines, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Willis Knighton Health System, Pierremont, Shreveport, Louisiana
  - Union Memorial Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Bay Regional Medical Center, Bay City, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Cooper Health System, Camden, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Gotham Cardiology, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Presbyterian Hospital - Charlotte, Charlotte, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pinnacle Health @ Harrisburg Hospital, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Northwest Texas Healthcare System, Amarillo, Texas
  - Heart Hospital of Austin, Austin, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital, Pearland, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Hospital, Bellingham, Washington
  - Heart Clinics Northwest/ Sacred Heart Medical Center, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (6):
  - Wesley Hospital, Auchenflower, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Monash Heart, Clayton, Victoria
  - St. Vincent's Hospital, Melbourne, Victoria
  - Epworth Hospital, Richmond, Victoria
  - Royal Perth Hospital, Perth, Western Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled into this trial will be male and female subjects from the general interventional cardiology population. The study commenced on June 5, 2009 with the first subject enrolled on June 15, 2009. The last subject in the CSR was enrolled February 12, 2010, and the last subject enrolled in LLR was on April 6, 2010.
Pre-assignment Details: Intention-to-treat (ITT) set includes 525 subjects: 415 in core size registry (CSR) arm and 110 in long lesion registry (LLR) arm. Full analysis set (FAS) (n=505, 401 in CSR arm and 104 in LLR arm) includes subjects who have received at least 1 of the following: the core size XIENCE PRIME or XIENCE PRIME LL stent system, including bailout.
Groups:
- Core Size Registry: Core size indicates the range of diameters of the stents used.
- Long Lesion Registry: Use of long lesion stents.
Period: Overall Study
Arm/Group | Core Size Registry | Long Lesion Registry
Started | 401 | 104
Completed | 396 | 102
Not Completed | 5 | 2
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data is presented for FAS population (n=505) for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Size Registry | Long Lesion Registry | Total
Number analyzed (Participants) | 401 | 104 | 505
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 234 | 56 | 290
  >=65 years | 167 | 48 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.70 (10.23) | 63.46 (9.44) | 62.86 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 39 | 158
  Male | 282 | 65 | 347
Region of Enrollment [Number; unit: participants]
  United States | 376 | 96 | 472
  Australia | 25 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure (TLF)
Description: The composite rate of:
  Cardiac Death Target Vessel Myocardial Infarction (TV-MI) and Clinically Indicated Target Lesion Revascularization (CI-TLR) per protocol.
Time Frame: 1 year
Population: The number of participants analyzed is based on FAS population, defined as subjects who have received the investigational study device and excludes subjects who are truly lost-to-follow-up, defined as subjects who are lost to follow-up through given timepoint without any DMR event (all death, all MI, all revascularization, respectively).
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 4.5 | 7.7

2. Secondary Outcome: Procedure Time
Description: Procedure time is defined as time between insertion and withdrawal of guide catheter.
Time Frame: From insertion to withdrawal of guide catheter
Population: The analysis was done to include only subjects with post index procedure cardiac enzyme data in window (between 8 hours post index procedure and hospital discharge). Therefore, the final analysis contained 403 ITT CSR subjects and 106 ITT LLR subjects.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 403 | 106
Minutes | 32.6 (21.1) | 46.9 (30.9)

3. Secondary Outcome: Device Success (Lesion Basis)
Description: Device success is defined as achievement of a final in-stent residual diameter stenosis of < 50% (by QCA).
Time Frame: From the start of index procedure to end of index procedure
Population: as for outcome 2
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 403 | 106
Number analyzed (Lesions) | 449 | 125
percentage of lesions | 98.2 | 97.6

4. Secondary Outcome: Procedural Success (Subject Basis)
Description: Procedure success is defined as achievement of a final in-stent diameter stenosis of < 50% (by QCA). Per Protocol.
Time Frame: From the start of index procedure to end of index procedure
Population: The analysis was done to include only subjects with post index procedure cardiac enzyme data in window (between 8 hours post index procedure and hospital discharge). Out of these subjects, 2 in the CSR and 1 in the LLR did not have QCA data and therefore were excluded. So, the final analysis contained 401 ITT CSR subjects and 105 ITT LLR subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 105
percentage of participants | 97.8 | 94.3

5. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Time Frame: In-hospital is less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.0 | 0.0

6. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.0 | 0.0

7. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 0.5 | 0.0

8. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 0.8 | 1.0

9. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 2.0 | 2.9

10. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 3.1 | 2.9

11. Secondary Outcome: Target Vessel-Myocardial Infarction (TV-MI) - Q-wave and Non Q-wave (Defined as MI Not Clearly Attributable to a Non-target Vessel)
Description: Per Protocol
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 1.7 | 4.8

12. Secondary Outcome: Target Vessel-Myocardial Infarction (TV-MI) - Q-wave and Non Q-wave (Defined as MI Not Clearly Attributable to a Non-target Vessel)
Description: Per Protocol
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 1.7 | 4.8

13. Secondary Outcome: Target Vessel-Myocardial Infarction (TV-MI) - Q-wave and Non Q-wave (Defined as MI Not Clearly Attributable to a Non-target Vessel)
Description: Per Protocol
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 1.8 | 4.8

14. Secondary Outcome: Target Vessel-Myocardial Infarction (TV-MI) - Q-wave and Non Q-wave (Defined as MI Not Clearly Attributable to a Non-target Vessel)
Description: Per Protocol
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 1.8 | 4.8

15. Secondary Outcome: Target Vessel-Myocardial Infarction (TV-MI) - Q-wave and Non Q-wave (Defined as MI Not Clearly Attributable to a Non-target Vessel)
Description: Per Protocol
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 1.8 | 4.8

16. Secondary Outcome: Target Vessel-Myocardial Infarction (TV-MI) - Q-wave and Non Q-wave (Defined as MI Not Clearly Attributable to a Non-target Vessel)
Description: Per Protocol
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 2.6 | 4.8

17. Secondary Outcome: Non-target Vessel MI (Q-wave, Non Q-wave)
Description: Per Protocol
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.0 | 0.0

18. Secondary Outcome: Non-target Vessel MI (Q-wave, Non Q-wave)
Description: Per Protocol
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.0 | 0.0

19. Secondary Outcome: Non-target Vessel MI (Q-wave, Non Q-wave)
Description: Per Protocol
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 0.0 | 0.0

20. Secondary Outcome: Non-target Vessel MI (Q-wave, Non Q-wave)
Description: Per Protocol
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 0.0 | 0.0

21. Secondary Outcome: Non-target Vessel MI (Q-wave, Non Q-wave)
Description: Per Protocol
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 0.3 | 1.9

22. Secondary Outcome: Non-target Vessel MI (Q-wave, Non Q-wave)
Description: Per Protocol
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 0.8 | 1.9

23. Secondary Outcome: Clinically Indicated-Target Lesion Revascularization
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.2 | 1.0

24. Secondary Outcome: Clinically Indicated-Target Lesion Revascularization
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.5 | 1.0

25. Secondary Outcome: Clinically Indicated-Target Lesion Revascularization
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 1.8 | 1.9

26. Secondary Outcome: Clinically Indicated-Target Lesion Revascularization
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 2.5 | 2.9

27. Secondary Outcome: Clinically Indicated-Target Lesion Revascularization
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 4.1 | 4.8

28. Secondary Outcome: Clinically Indicated-Target Lesion Revascularization
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 5.4 | 4.8

29. Secondary Outcome: Clinically Indicated Target Vessel Revascularization (TVR = TLR and Non-TLR in TV)
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.5 | 1.0

30. Secondary Outcome: Clinically Indicated Target Vessel Revascularization (TVR = TLR and Non-TLR in TV)
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 1.2 | 1.9

31. Secondary Outcome: Clinically Indicated Target Vessel Revascularization (TVR = TLR and Non-TLR in TV)
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 3.3 | 3.8

32. Secondary Outcome: Clinically Indicated Target Vessel Revascularization (TVR = TLR and Non-TLR in TV)
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 4.5 | 4.8

33. Secondary Outcome: Clinically Indicated Target Vessel Revascularization (TVR = TLR and Non-TLR in TV)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 6.9 | 7.7

34. Secondary Outcome: Clinically Indicated Target Vessel Revascularization (TVR = TLR and Non-TLR in TV)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 9.5 | 7.7

35. Secondary Outcome: All TLR (CI and Non-CI)
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.2 | 1.0

36. Secondary Outcome: All TLR (CI and Non-CI)
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.5 | 1.0

37. Secondary Outcome: All TLR (CI and Non-CI)
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 2.0 | 1.9

38. Secondary Outcome: All TLR (CI and Non-CI)
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 2.8 | 2.9

39. Secondary Outcome: All TLR (CI and Non-CI)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 4.3 | 4.8

40. Secondary Outcome: All TLR (CI and Non-CI)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 5.6 | 4.8

41. Secondary Outcome: All TVR (CI and Non-CI)
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.5 | 1.0

42. Secondary Outcome: All TVR (CI and Non-CI)
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 1.2 | 1.9

43. Secondary Outcome: All TVR (CI and Non-CI)
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 3.5 | 3.8

44. Secondary Outcome: All TVR (CI and Non-CI)
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 4.8 | 4.8

45. Secondary Outcome: All TVR (CI and Non-CI)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 7.1 | 7.7

46. Secondary Outcome: All TVR (CI and Non-CI)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 10 | 7.7

47. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 0.5 | 1.0

48. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 1.5 | 3.8

49. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 4.8 | 6.7

50. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 6.8 | 8.7

51. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 10.5 | 13.5

52. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 14.9 | 14.4

53. Secondary Outcome: Cardiac Death/All MI
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 1.7 | 4.8

54. Secondary Outcome: Cardiac Death/ All MI
Description: Per Protocol
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 1.7 | 4.8

55. Secondary Outcome: Cardiac Death/All MI
Description: Per Protocol
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 2.0 | 4.8

56. Secondary Outcome: Cardiac Death/All MI
Description: Per Protocol
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 2.0 | 4.8

57. Secondary Outcome: Cardiac Death/All MI
Description: Per Protocol
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 2.6 | 5.8

58. Secondary Outcome: Cardiac Death/All MI
Description: Per Protocol
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 3.8 | 5.8

59. Secondary Outcome: Cardiac Death/ All MI/CI-TLR
Time Frame: in-hospital
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 2.0 | 5.8

60. Secondary Outcome: Cardiac Death/ All MI/CI-TLR
Description: Per Protocol
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 2.2 | 5.8

61. Secondary Outcome: Cardiac Death/ All MI/CI-TLR
Description: Per Protocol
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 3.8 | 6.7

62. Secondary Outcome: Cardiac Death/ All MI/CI-TLR
Description: Per Protocol
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 4.5 | 7.7

63. Secondary Outcome: Cardiac Death/ All MI/CI-TLR
Description: Per Protocol
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 6.6 | 10.6

64. Secondary Outcome: Cardiac Death/ All MI/CI-TLR
Description: Per Protocol
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 9.0 | 10.6

65. Secondary Outcome: All Death/All MI/All Coronary Revascularization
Description: Per Protocol
Time Frame: In-hospital is defined as hospitalization less than or equal to 7 days post index procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 2.2 | 5.8

66. Secondary Outcome: All Death/All MI/All Coronary Revascularization
Description: Per Protocol
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants | 3.2 | 8.7

67. Secondary Outcome: All Death/All MI/All Coronary Revascularization
Description: Per Protocol
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 7.0 | 11.5

68. Secondary Outcome: All Death/All MI/All Coronary Revascularization
Description: Per Protocol
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants | 9.0 | 14.4

69. Secondary Outcome: All Death/All MI/All Coronary Revascularization
Description: Per Protocol
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 13.8 | 20.2

70. Secondary Outcome: All Death/All MI/All Coronary Revascularization
Description: Per Protocol
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 19 | 20.2

71. Secondary Outcome: Stent Thrombosis
Description: Per protocol and per Academic Research Consortium (ARC, definite/probable)
Time Frame: Acute (≤1 day)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants
  Per ARC | 0.5 | 0.0
  Per Protocol | 0.5 | 0.0

72. Secondary Outcome: Stent Thrombosis
Description: Per protocol and per ARC
Time Frame: Subacute (>1 - 30 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants
  Per ARC | 0.0 | 0.0
  Per Protocol | 0.0 | 0.0

73. Secondary Outcome: Stent Thrombosis
Description: Per protocol and per ARC
Time Frame: Acute/Subacute (0 - 30 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 401 | 104
percentage of participants
  Per ARC | 0.5 | 0.0
  Per Protocol | 0.5 | 0.0

74. Secondary Outcome: Stent Thrombosis
Description: Per protocol and per ARC
Time Frame: Late (31 - 393 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants
  Per ARC | 0.0 | 0.0
  Per Protocol | 0.0 | 0.0

75. Secondary Outcome: Stent Thrombosis
Description: Per protocol
Time Frame: Late (31 - 758 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 385 | 100
percentage of participants | 0.3 | 0.0

76. Secondary Outcome: Stent Thrombosis
Description: Per ARC, definite and probable
Time Frame: Very Late (394 - 758 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 385 | 100
percentage of participants | 0.0 | 0.0

77. Secondary Outcome: Stent Thrombosis
Description: Per protocol
Time Frame: Late (31 - 1123 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 378 | 99
percentage of participants | 0.5 | 0.0

78. Secondary Outcome: Stent Thrombosis
Description: Per ARC, definite and probable
Time Frame: Very Late (394 - 1123 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 379 | 99
percentage of participants | 0.3 | 0

79. Primary Outcome: Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 392 | 104
percentage of participants | 6.4 | 9.6

80. Primary Outcome: Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 390 | 104
percentage of participants | 8.5 | 9.6

81. Secondary Outcome: Stent Thrombosis
Description: Per protocol and per ARC
Time Frame: Overall (0-393 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 399 | 104
percentage of participants
  Per ARC | 0.5 | 0.0
  Per Protocol | 0.5 | 0.0

82. Secondary Outcome: Stent Thrombosis
Description: Per protocol
Time Frame: Overall (0-758 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 385 | 100
percentage of participants | 0.8 | 0.0

83. Secondary Outcome: Stent Thrombosis
Description: Per ARC, definite and probable
Time Frame: Overall (0-758 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 386 | 100
percentage of participants | 0.5 | 0

84. Secondary Outcome: Stent Thrombosis
Description: Per protocol
Time Frame: Overall (0 - 1123 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 378 | 99
percentage of participants | 1.1 | 0.0

85. Secondary Outcome: Stent Thrombosis
Description: Per ARC, definite and probable
Time Frame: Overall (0 - 1123 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Size Registry | Long Lesion Registry
Number analyzed (Participants) | 380 | 99
percentage of participants | 0.8 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: These are site-reported, un-adjudicated adverse events regardless of relationship to the device in intention-to-treat population. The number of participants at risk excludes subjects who were early terminated up to 1123 days and had no events through the given timepoint
Arm/Group | Core Size Registry | Long Lesion Registry
Serious Adverse Events (participants affected / at risk) | 203/412 | 49/110
Other Adverse Events (participants affected / at risk) | 222/412 | 51/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Size Registry (N=412) | Long Lesion Registry (N=110)
Acute myocardial infarction (Cardiac disorders) | 12 (13) | 3 (4)
Angina pectoris (Cardiac disorders) | 59 (83) | 16 (20)
Angina unstable (Cardiac disorders) | 14 (21) | 6 (6)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 9 (10) | 2 (2)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 8 (10) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 7 (8) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 3 (3) | 2 (2)
Coronary artery embolism (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 4 (4) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (3) | 0 (0)
Microvascular angina (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Post procedural myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 23 (30) | 6 (6)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lead dislodgement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombosis in device (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Other injuries (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) — Other injuries consists of all the Preferred Terms (PT) which were not in Administration site reactions and Procedural and device related injuries and classifications High-Level Group Terms category for the corresponding System Organ Class (SOC)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (2)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 7 (8) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo positional (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Other renal and urinary disorders (Renal and urinary disorders) | 6 (7) | 3 (3) — Other renal and urinary disorders consist of all the PTs which were not in Acute renal failure for the corresponding SOC.
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wegeners granulomatosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 3 (4) | 0 (0)
Carotid artery stenosis (Vascular disorders) | 4 (4) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 0 (0)
Duodenal ulcer haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Epistaxis (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 2 (3)
Gastrointestinal haemorrhage (Vascular disorders) | 3 (3) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemoptysis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (2)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 2 (2)
Post procedural haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 2 (2) | 0 (0)
Scrotal haematocoele (Vascular disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Subdural haematoma (Vascular disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barretts oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Exomphalos (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (3)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (2)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Serratia infection (Infections and infestations) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 3 (3) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Pedal pulse decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (11) | 5 (6)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Intentional overdose (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 3 (3) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (2) | 0 (0)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Size Registry (N=412) | Long Lesion Registry (N=110)
Angina pectoris (Cardiac disorders) | 89 (114) | 20 (24)
Coronary artery dissection (Cardiac disorders) | 11 (11) | 9 (9)
Catheter site haematoma (General disorders) | 21 (21) | 5 (5)
Fatigue (General disorders) | 25 (25) | 3 (3)
Non-cardiac chest pain (General disorders) | 71 (77) | 13 (14)
Headache (Nervous system disorders) | 27 (27) | 3 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (27) | 3 (3)
Hypertension (Vascular disorders) | 11 (12) | 6 (6)
Catheter site haemorrhage (General disorders) | 15 (16) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (28) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication except to delay any proposed publication or presentation to enable the Sponsor to secure patent or other protection of proprietary rights.